CLINICAL TRIAL: NCT02697084
Title: Individual Following in Anal Cancer With PET/CT
Acronym: IFACT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/54
Record Dates: First submitted 2016-02-22; First posted 2016-03-03 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Anal Cancer
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: anal cancer — Anal cancer patients with TEP TDM

SUMMARY:
Anal canal cancer is a relatively rare disease, representing 1.2% of digestive cancers and 6% of anorectal cancers. Incidence is less than 1/100 000 of the general population. However, the incidence has increased considerably over the past three decades. The main risk factors are HPV infections and smoking. Initial treatment comprises radiochemotherapy or radiotherapy alone, according to the patient's tumor stage and tolerance of chemotherapy. The choice of the most appropriate treatment strategy will condition the patient's prognosis. Consequently, early assessment of the initial extension of the tumor, its therapeutic response and relapses constitute determining factors in the management of the disease Despite the good results obtained, persistent disease is observed in 30% of cases and abdominal-pelvic salvage amputation can then prove effective in cases of local or loco-regional relapse. The great majority of relapses occur within 2 years after treatment. Reported prognostic survival factors are the T stage, size inferior or superior to 4 cm and inguinal or pelvic lymph node involvement.

The rules for follow-up are not substantiated by high levels of proof. Follow-up focuses principally on the clinical examination although the type and frequency of the paraclinical examinations are not backed by any consensus.

DETAILED DESCRIPTION:
Post-treatment 18-FDG PET scan at 2 months can prove useful to predict locoregional or metastatic recurrence in patients treated by radiochemotherapy or radiotherapy in the anal canal cancer setting. There appear to be an FDG intensity variable and a metabolic response criterion enabling establishment of two groups of patients: low recurrence risk versus high recurrence risk at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive inclusion of incident cases of anal canal cancer between November 2014 and May 2018. These patients are volunteers and have signed informed consent.

Exclusion Criteria:

* Presence of a nother cancer and specific treatment (chemotherapy, radiotherapy). Follow-up impossible during two years or more.

Refusal to submit to initial or post-treatment PET/CT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Canal anal cancer
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2014-11; Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
time of disease-free survival | 3 years

SECONDARY OUTCOMES:
best metabolic response measurement variable: SUVmax | 3 years
best metabolic response measurement variable: SUVmean | 3 years
best metabolic response measurement variable: SUL peak | 3 years
best metabolic response measurement variable: Metabolic Total Volume (MTV) | 3 years
best metabolic response measurement variable: Total Lesion Glycolysis (TLG) | 3 years
best treatment response criterion: SUV or metabolic volume threshold | 3 years
best treatment response criterion: ratio (SUV or metabolic volume) | 3 years
best treatment response criterion: complete or partial metabolic response according to EORTC or PERCIST criteria | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: LOVERA Christine, Study Director — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: No